CLINICAL TRIAL: NCT05840913
Title: Comparison of Anaesthetic Effectiveness of Different Volumes of Articaine for Inferior Alveolar Nerve Block in Molar Teeth with Symptomatic Irreversible Pulpitis
Brief Title: Different Volumes of Articaine for Inferior Alveolar Nerve Block in Irreversible Pulpitis
Acronym: IANB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Kanza Zafar, Dr. Kanza Zafar, Principal Investigator and Resident Operative Dentistry and Endodontics, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Articaine Efficacy for IANB
Record Dates: First submitted 2023-04-09; First posted 2023-05-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Drug Effect; Pulpitis - Irreversible
MeSH Terms: interventions — Carticaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1.8 ml group (Experimental): Participants in this group will be given 1 cartridge of articaine solution pre-operatively to endodontic treatment
  Interventions: Drug: Articaine HCl 4 % / EPINEPHrine 1:100,000 in 1.8 mL Dental Cartridge
- 3.6 ml group (Experimental): Participants in this group will be given 2 cartridges of articaine solution pre-operatively to endodontic treatment
  Interventions: Drug: Articaine HCl 4 % / EPINEPHrine 1:100,000 in 1.8 mL Dental Cartridge

INTERVENTIONS:
Drug: Articaine HCl 4 % / EPINEPHrine 1:100,000 in 1.8 mL Dental Cartridge — Local anesthetic injection for intra- operative pain control
  Other Names: Orabloc 4% Articaine 1:100,000 1.8 ml

SUMMARY:
This is a randomized controlled trial comparing the anaesthetic efficacy of 1.8 and 3.6 mL of Articaine for inferior alveolar nerve block when treating mandibular molars with Irreversible Pulpitis

DETAILED DESCRIPTION:
An informed written consent of the patients will be obtained. (Annex-A).

Demographic details (including name, age, gender, contact) will be obtained on data collection forms. (Annex-B).

The principal investigator will perform the local anesthetic injection and the participants will be assigned to one of the groups.

Group 1: 1.8 mL articaine Group 2: 3.6 mL articaine

Before starting the treatment i.e. before administration of the anesthetic solution, each participant will receive an explanation regarding the Heft-Parker visual analog pain scale (VAS) and asked to rate their pain on a self-report questionnaire.

A topical anesthetic gel (20% Benzocaine; Premier, Philadelphia, PA) will passively placed at the injection site with a cotton tip applicator for 1 minute before injection.

A conventional IANB will administered using an aspirating syringe with a side-loading cartridge system (Dena Instruments; Forgeman Instruments Co, Sialkot, Pakistan) and a 27-G 31-mm needle (C-K ject; CK Dental, Kor-Kyungji-do, Korea).

All injections will be given by one clinician in both groups. Group 2 participants will receive 2 cartridges of the anesthetic solution and group 1 will receive a cartridge of the anesthetic solution followed by a mock injection.

The rest of the procedure will be performed by a second investigator. Ten minutes after injection, the participants will be asked whether they have lip numbness. Any patient without lip numbness at this stage will excluded from study.

Fifteen minutes after the administration of the IANB, the teeth will be re-evaluated with electric pulp testing. On positive response, participants will be again asked to rate their pain using the VAS on the questionnaire.

If higher than mild pain is reported, supplemental anesthesia (intraperiodontal ligament or intrapulpal injection) will be used to provide patient comfort throughout the treatment.

Then teeth under study will be isolated with a rubber dam, and caries removed followed by the preparation of an endodontic access cavity. The participants will be informed to stop the practitioner at any stage of treatment if they feel more than mild pain by raising their hand.

At the end of each stage of treatment (access cavity preparation, pulp chamber opening, root canal instrumentation), the practitioner will stop work and ask the participants to rate their pain if they do not raise their hand during treatment.

The success will be defined as the ability to undertake pulp access and canal instrumentation with no or mild pain whereas moderate or severe pain will considered as failure of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients, including age group 18-55 years old
* Mandibular first molar tooth with symptomatic irreversible pulpitis
* Normal periapical radiographic appearance
* Moderate pain on Heft-Parker VAS ( > 54 mm and < 114 mm )
* Lingering pain or prolonged response to the cold testing (more than 10 seconds)
* Positive response to electric pulp testing

Exclusion Criteria:

* Patients who have taken analgesic or anti-inflammatory drugs within 6 hours before treatment visit
* History of allergy to 4% articaine or epinephrine
* Patients with systemic diseases
* Pregnant or lactating patients
* Teeth with severe periodontal disease
* Teeth with periapical radiolucency
* Any type of medication that could potentially interact with the anesthetic solution (antihypertensives)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Pain Control | 30 to 45 minutes
  Pain was recorded on a self-report questionnaire using the visual analog pain scale (VAS) VAS was used for gauging pain before the administration of the anesthetic solution, after the cold test was performed, and during the endodontic therapy.
  The VAS scores were designated as; 0= no pain 1-3= mild pain 4-7= moderate pain 8-10= severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Kanza Zafar, BDS, Principal Investigator — AFID
Locations (2):
- Pakistan (2):
  - Armed Forces Institue Of Dentistry, Rawalpindi, Punjab Province
  - Armed Forces Institute of Dentistry, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No